CLINICAL TRIAL: NCT00715481
Title: Reduced Estimated Glomerular Filtration Rate (eGFR)and Prediction of Cardiovascular Disease and Renal Outcome in Subjects With Type 2 Diabetes: Italian Multicenter Study
Brief Title: Renal Insufficiency And Cardiovascular Events
Acronym: RIACE
Status: Completed | Type: Observational
Sponsor: Diabetic Nephropathy Study Group (Other)
Collaborators: Italian Society of Diabetology (Other)
Responsible Party: Principal Investigator, Giuseppe Pugliese, Professor of Endocrinology and Metabolism, Diabetic Nephropathy Study Group
Other Study IDs: DNSG-SID 0601
Record Dates: First submitted 2008-07-10; First posted 2008-07-15 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Cardiovascular Disease
Keywords: Type 2 diabetes; Cardiovascular disease; Diabetic Nephropathy; Glomerular filtration rate; Albuminuria
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus, Type 2; Diabetic Nephropathies; Albuminuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Reduced glomerular filtration rate (GFR) has been recently shown to be a powerful predictor of cardiovascular morbidity and mortality in the general population, independent of traditional cardiovascular risk factors.

This observational study is aimed at assessing the association of reduced estimated GFR with cardiovascular morbidity and mortality in a large italian population (at least 15,000 subjects) of type 2 diabetic outpatients over a 4-year follow-up.

DETAILED DESCRIPTION:
Reduced GFR has been recently shown to be a powerful predictor of cardiovascular morbidity and mortality in the general population, independent of traditional cardiovascular risk factors. Since type 2 diabetic patients show increased cardiovascular morbidity and mortality as compared with the general population, the identification of predictors of cardiovascular disease in these patients is of fundamental importance for clinical purposes. One of these predictors is increased urinary albumin excretion rate, which is associated with an increased risk of cardiovascular disease more than of end-stage renal disease. However, a growing body of evidence indicates that a significant proportion of normoalbuminuric diabetic patients, particularly with type 2 diabetes, may exhibit reduced GFR. It is currently unknown the predictive role of this abnormality toward cardiovascular events and death, independent of albuminuria and other known risk factors, in the diabetic population.

This observational study is aimed at assessing the association of reduced estimated GFR with cardiovascular morbidity and mortality in a large italian population (at least 15,000 subjects) of type 2 diabetic nondialytic outpatients over a 4-year follow-up.

Secondary endpoints are to assess in this population:

* the prevalence and incidence of reduced GFR, as classified according to the National Kidney Foundation criteria, and its association with traditional cardiovascular risk factors;
* the prevalence, incidence and cardiovascular predictivity of micro and macroalbuminuria.

Patients will be recruited from electronic records of 20 italian outpatients diabetic clinics.

Routine anamnestic, clinical, laboratory and instrumental data will be recorded at baseline and over 4 years to obtain information about:

* renal function (albumin/creatinine ratio, serum creatinine with estimation of glomerular filtration rate [eGFR]);
* cardiovascular risk factors (smoking, physical activity, family history of diabetes, dyslipidemia, hypertension and cardiovascular disease, BMI and waist circumference, total, LDL, HDL and non-HDL cholesterol, triglycerides, arterial blood pressure and HbA1c);
* current glucose-, lipid- and blood pressure-lowering and anti-platelet or anti-coagulant treatment;
* other illnesses;
* cardiovascular events (myocardial infarction, stroke, lower limb ulcer/gangrene/amputation and coronary, carotid and lower limb revascularization, endovascular/surgical) and deaths.

These data will be derived from the electronic database of each participating center.

Laboratory analyses will be performed in each centre laboratory after proper standardization of analytical techniques.

ELIGIBILITY:
Inclusion Criteria:

type 2 diabetes

Exclusion Criteria:

dyalisis or renal transplantation

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients clinics
Sampling Method: Probability Sample
Enrollment: 15628 (Actual)
Dates: Start 2008-06; Primary Completion 2008-11 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
cardiovascular morbidity and mortality | 4 years

SECONDARY OUTCOMES:
eGFR, as classified according to the National Kidney Foundation criteria | 4 years
micro/macroalbuminuria | 4 years
traditional cardiovascular risk factors | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Pugliese, MD, PhD, Principal Investigator — Diabetic Nephropathy Study Group; Anna Solini, MD, PhD, Study Director — Diabetic Nephropathy Study Group
Locations (20):
- Italy (20):
  - Mazzoni Hospital, Division of Diabetology, Ascoli Piceno
  - Policlinico Hospital, Division of Endocrinology, Bari
  - Ospedali Riuniti di Bergamo, Division of Diabetology, Bergamo
  - Monserrato Hospital, Division of Diabetology, Cagliari
  - Mater Domini Hospital, Division of Internal Medicine, Catanzaro
  - Policlinico Hospital, Division of Endocrinology, Foggia
  - Santa Maria Goretti Hospital, Division of Diabetology, Latina
  - Policlinico - Maggiore Hospital, Division of Endocrinology and Diabetology, Milan
  - San Giuseppe Hospital, Division of Endocrinology, Milan
  - San Raffaele Hospital, Milan
  - San Paolo Hospital, Division of Internal Medicine, Milan
  - San Luigi Gonzaga Hospital, Division of Diabetes and Metabolic Diseases, Orbassano-Torino
  - Policlinico Hospital, Division of Diabetology, Padua
  - Cisanello Hospital, Divisions of Diabetology, Pisa
  - Santa Chiara Hospital, Division of Internal Medicine, Pisa
  - Policlinico Hospital, Division of Internal Medicine, Rome
  - Sant'Andrea Hospital, Division of Diabetology, Rome
  - Policlinico Le Scotte, Division of Diabetology, Siena
  - Le Molinette - San Giovanni Battista Hospital, Division of Diabetology, Torino
  - Maggiore Hospital, Division of Endocrinology and Metabolic Diseases, Verona

REFERENCES:
- [Derived] Garofolo M, Penno G, Solini A, Orsi E, Vitale M, Resi V, Bonora E, Fondelli C, Trevisan R, Vedovato M, Nicolucci A, Pugliese G; Renal Insufficiency And Cariovascular Events (RIACE) Study Group. Association of Albuminuria Within the Normoalbuminuric Range With All-Cause Mortality in People With Type 2 Diabetes. Diabetes Metab Res Rev. 2025 Jul;41(5):e70061. doi: 10.1002/dmrr.70061. PMID 40557728
- [Derived] Garofolo M, Vitale M, Penno G, Solini A, Orsi E, Grancini V, Bonora E, Fondelli C, Trevisan R, Vedovato M, Nicolucci A, Pugliese G; Renal Insufficiency And Cardiovascular Events (RIACE) Study Group. Prognostic impact of switching to the 2021 chronic kidney disease epidemiology collaboration creatinine-based equation in Caucasian patients with type 2 diabetes: the Renal Insufficiency and Cardiovascular events (RIACE) Italian Multicenter Study. Cardiovasc Diabetol. 2024 Oct 24;23(1):377. doi: 10.1186/s12933-024-02450-5. PMID 39449120
- [Derived] Garofolo M, Penno G, Solini A, Orsi E, Vitale M, Resi V, Bonora E, Fondelli C, Trevisan R, Vedovato M, Nicolucci A, Pugliese G; Renal Insufficiency And Cardiovascular Events (RIACE) Study Group. Relationship between degree of risk factor control and all-cause mortality in individuals with type 2 diabetes: A prospective cohort study. Eur J Intern Med. 2024 Oct;128:53-62. doi: 10.1016/j.ejim.2024.05.034. Epub 2024 Jun 6. PMID 38845288
- [Derived] Vitale M, Orsi E, Solini A, Garofolo M, Grancini V, Bonora E, Fondelli C, Trevisan R, Vedovato M, Penno G, Nicolucci A, Pugliese G; Renal Insufficiency And Cardiovascular Events (RIACE) Study Group*. Association between age at diagnosis and all-cause mortality in type 2 diabetes: the Renal Insufficiency and Cardiovascular Events (RIACE) Italian Multicenter Study. Acta Diabetol. 2024 Sep;61(9):1107-1116. doi: 10.1007/s00592-024-02294-1. Epub 2024 May 7. PMID 38714557
- [Derived] Vitale M, Orsi E, Solini A, Garofolo M, Resi V, Bonora E, Fondelli C, Trevisan R, Vedovato M, Penno G, Pugliese G. Independent association of history of diabetic foot with all-cause mortality in patients with type 2 diabetes: the Renal Insufficiency And Cardiovascular Events (RIACE) Italian Multicenter Study. Cardiovasc Diabetol. 2024 Jan 13;23(1):34. doi: 10.1186/s12933-023-02107-9. PMID 38218843
- [Derived] Solini A, Orsi E, Vitale M, Garofolo M, Resi V, Bonora E, Fondelli C, Trevisan R, Vedovato M, Nicolucci A, Penno G, Pugliese G; Renal Insufficiency And Cardiovascular Events (RIACE) Study Group. Independent association of estimated pulse-wave velocity with all-cause mortality in individuals with type 2 diabetes. QJM. 2024 Jul 1;117(7):495-502. doi: 10.1093/qjmed/hcae012. PMID 38200621
- [Derived] Orsi E, Solini A, Penno G, Bonora E, Fondelli C, Trevisan R, Vedovato M, Cavalot F, Lamacchia O, Haxhi J, Nicolucci A, Pugliese G; Renal Insufficiency And Cardiovascular Events (RIACE) Study Group. Body mass index versus surrogate measures of central adiposity as independent predictors of mortality in type 2 diabetes. Cardiovasc Diabetol. 2022 Dec 2;21(1):266. doi: 10.1186/s12933-022-01706-2. PMID 36461034
- [Derived] Orsi E, Solini A, Bonora E, Vitale M, Garofolo M, Fondelli C, Trevisan R, Vedovato M, Cavalot F, Laviola L, Morano S, Pugliese G; Renal Insufficiency And Cardiovascular Events (RIACE) Study Group. Risk of all-cause mortality according to the European Society of Cardiology risk categories in individuals with type 2 diabetes: the Renal Insufficiency And Cardiovascular Events (RIACE) Italian Multicenter Study. Acta Diabetol. 2022 Oct;59(10):1369-1381. doi: 10.1007/s00592-022-01942-8. Epub 2022 Jul 28. PMID 35902419
- [Derived] Penno G, Solini A, Orsi E, Bonora E, Fondelli C, Trevisan R, Vedovato M, Cavalot F, Zerbini G, Lamacchia O, Nicolucci A, Pugliese G; Renal Insufficiency And Cardiovascular Events (RIACE) Study Group. Insulin resistance, diabetic kidney disease, and all-cause mortality in individuals with type 2 diabetes: a prospective cohort study. BMC Med. 2021 Mar 15;19(1):66. doi: 10.1186/s12916-021-01936-3. PMID 33715620
- [Derived] Orsi E, Penno G, Solini A, Bonora E, Fondelli C, Trevisan R, Vedovato M, Cavalot F, Morano S, Baroni MG, Nicolucci A, Pugliese G; Renal Insufficiency And Cardiovascular Events (RIACE) Study Group. Independent association of atherogenic dyslipidaemia with all-cause mortality in individuals with type 2 diabetes and modifying effect of gender: a prospective cohort study. Cardiovasc Diabetol. 2021 Jan 30;20(1):28. doi: 10.1186/s12933-021-01224-7. PMID 33516215
- [Derived] Penno G, Orsi E, Solini A, Bonora E, Fondelli C, Trevisan R, Vedovato M, Cavalot F, Gruden G, Laviola L, Nicolucci A, Pugliese G; Renal Insufficiency And Cardiovascular Events (RIACE) Study Group. Renal hyperfiltration is independently associated with increased all-cause mortality in individuals with type 2 diabetes: a prospective cohort study. BMJ Open Diabetes Res Care. 2020 Jul;8(1):e001481. doi: 10.1136/bmjdrc-2020-001481. PMID 32665314
- [Derived] Solini A, Penno G, Orsi E, Bonora E, Fondelli C, Trevisan R, Vedovato M, Cavalot F, Lamacchia O, Baroni MG, Nicolucci A, Pugliese G; Renal Insufficiency And Cardiovascular Events (RIACE) Study Group. Is resistant hypertension an independent predictor of all-cause mortality in individuals with type 2 diabetes? A prospective cohort study. BMC Med. 2019 Apr 25;17(1):83. doi: 10.1186/s12916-019-1313-x. PMID 31023377
- [Derived] Penno G, Solini A, Orsi E, Bonora E, Fondelli C, Trevisan R, Vedovato M, Cavalot F, Lamacchia O, Scardapane M, Nicolucci A, Pugliese G; Renal Insufficiency And Cardiovascular Events (RIACE) Study Group. Non-albuminuric renal impairment is a strong predictor of mortality in individuals with type 2 diabetes: the Renal Insufficiency And Cardiovascular Events (RIACE) Italian multicentre study. Diabetologia. 2018 Nov;61(11):2277-2289. doi: 10.1007/s00125-018-4691-2. Epub 2018 Jul 21. PMID 30032426
- [Derived] Penno G, Solini A, Bonora E, Orsi E, Fondelli C, Zerbini G, Trevisan R, Vedovato M, Cavalot F, Laviola L, Nicolucci A, Pugliese G; Renal Insufficiency and Cardiovascular Events (RIACE) Study Group. Defining the contribution of chronic kidney disease to all-cause mortality in patients with type 2 diabetes: the Renal Insufficiency And Cardiovascular Events (RIACE) Italian Multicenter Study. Acta Diabetol. 2018 Jun;55(6):603-612. doi: 10.1007/s00592-018-1133-z. Epub 2018 Mar 24. PMID 29574497
- [Derived] Penno G, Solini A, Zoppini G, Fondelli C, Trevisan R, Vedovato M, Cavalot F, Gruden G, Lamacchia O, Laviola L, Orsi E, Pugliese G; Renal Insufficiency Cardiovascular Events (RIACE) Study Group. Independent correlates of urinary albumin excretion within the normoalbuminuric range in patients with type 2 diabetes: The Renal Insufficiency And Cardiovascular Events (RIACE) Italian Multicentre Study. Acta Diabetol. 2015 Oct;52(5):971-81. doi: 10.1007/s00592-015-0789-x. Epub 2015 Jul 10. PMID 26155957
- [Derived] Penno G, Solini A, Zoppini G, Fondelli C, Trevisan R, Vedovato M, Gruden G, Lamacchia O, Pontiroli AE, Arosio M, Orsi E, Pugliese G; Renal Insufficiency And Cardiovascular Events (RIACE) Study Group. Hypertriglyceridemia Is Independently Associated with Renal, but Not Retinal Complications in Subjects with Type 2 Diabetes: A Cross-Sectional Analysis of the Renal Insufficiency And Cardiovascular Events (RIACE) Italian Multicenter Study. PLoS One. 2015 May 5;10(5):e0125512. doi: 10.1371/journal.pone.0125512. eCollection 2015. PMID 25942403
- [Derived] Pugliese G, Solini A, Bonora E, Orsi E, Zerbini G, Fondelli C, Gruden G, Cavalot F, Lamacchia O, Trevisan R, Vedovato M, Penno G; RIACE Study Group. Distribution of cardiovascular disease and retinopathy in patients with type 2 diabetes according to different classification systems for chronic kidney disease: a cross-sectional analysis of the renal insufficiency and cardiovascular events (RIACE) Italian multicenter study. Cardiovasc Diabetol. 2014 Mar 13;13:59. doi: 10.1186/1475-2840-13-59. PMID 24624891
- [Derived] Penno G, Solini A, Zoppini G, Orsi E, Fondelli C, Zerbini G, Morano S, Cavalot F, Lamacchia O, Trevisan R, Vedovato M, Pugliese G; Renal Insufficiency and Cardiovascular Events (RIACE) Study Group. Hemoglobin A1c variability as an independent correlate of cardiovascular disease in patients with type 2 diabetes: a cross-sectional analysis of the renal insufficiency and cardiovascular events (RIACE) Italian multicenter study. Cardiovasc Diabetol. 2013 Jul 5;12:98. doi: 10.1186/1475-2840-12-98. PMID 23829205
- [Derived] Penno G, Solini A, Bonora E, Fondelli C, Orsi E, Zerbini G, Trevisan R, Vedovato M, Gruden G, Laviola L, Nicolucci A, Pugliese G; Renal Insufficiency And Cardiovascular Events (RIACE) study, group. Gender differences in cardiovascular disease risk factors, treatments and complications in patients with type 2 diabetes: the RIACE Italian multicentre study. J Intern Med. 2013 Aug;274(2):176-91. doi: 10.1111/joim.12073. Epub 2013 Apr 22. PMID 23565931
- [Derived] Penno G, Solini A, Bonora E, Fondelli C, Orsi E, Zerbini G, Morano S, Cavalot F, Lamacchia O, Laviola L, Nicolucci A, Pugliese G; Renal Insufficiency And Cardiovascular Events Study Group. HbA1c variability as an independent correlate of nephropathy, but not retinopathy, in patients with type 2 diabetes: the Renal Insufficiency And Cardiovascular Events (RIACE) Italian multicenter study. Diabetes Care. 2013 Aug;36(8):2301-10. doi: 10.2337/dc12-2264. Epub 2013 Mar 14. PMID 23491522
- [Derived] Penno G, Solini A, Zoppini G, Orsi E, Zerbini G, Trevisan R, Gruden G, Cavalot F, Laviola L, Morano S, Nicolucci A, Pugliese G; Renal Insufficiency And Cardiovascular Events (RIACE) Study Group. Rate and determinants of association between advanced retinopathy and chronic kidney disease in patients with type 2 diabetes: the Renal Insufficiency And Cardiovascular Events (RIACE) Italian multicenter study. Diabetes Care. 2012 Nov;35(11):2317-23. doi: 10.2337/dc12-0628. PMID 23093684
- [Derived] Pugliese G, Solini A, Zoppini G, Fondelli C, Zerbini G, Vedovato M, Cavalot F, Lamacchia O, Buzzetti R, Morano S, Nicolucci A, Penno G; Renal Insufficiency and Cardiovascular Events (RIACE) Study Group. High prevalence of advanced retinopathy in patients with type 2 diabetes from the Renal Insufficiency And Cardiovascular Events (RIACE) Italian Multicenter Study. Diabetes Res Clin Pract. 2012 Nov;98(2):329-37. doi: 10.1016/j.diabres.2012.09.006. Epub 2012 Sep 26. PMID 23020932
- [Derived] Pugliese G, Solini A, Fondelli C, Trevisan R, Vedovato M, Nicolucci A, Penno G; Renal Insufficiency And Cardiovascular Events (RIACE) Study Group. Reproducibility of albuminuria in type 2 diabetic subjects. Findings from the Renal Insufficiency And Cardiovascular Events (RIACE) study. Nephrol Dial Transplant. 2011 Dec;26(12):3950-4. doi: 10.1093/ndt/gfr140. Epub 2011 Mar 25. PMID 21441399